CLINICAL TRIAL: NCT06003673
Title: A Single-arm Exploratory Clinical Study of Tislelizumab Combined With Transarterial Chemoembolization (TACE) and Lenvatinib in the Neoadjuvant Treatment of Resectable CNLC Stage Ⅱa-Ⅱb Hepatocellular Carcinoma
Brief Title: A Clinical Study of Tislelizumab Combined With TACE and Lenvatinib in the Neoadjuvant Treatment of Resectable HCC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Zhang Zhibo, Director of Hepatobiliary and Pancreatic Surgery Department, First Affiliated Hospital of Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRCTA.ECFAH of FMU[2023]405
Record Dates: First submitted 2023-08-14; First posted 2023-08-22 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Hepatocellular Carcinoma Resectable
Keywords: hepatocellular carcinoma; resectable; CNLC stage IIa-IIb; neoadjuvant therapy; Tislelizumab; Lenvatinib; Transarterial Chemoembolization (TACE)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant therapy group (Experimental): Participants will receive a combination treatment of Tislelizumab, Lenvatinib, and Transarterial Chemoembolization (TACE).
  Interventions: Combination Product: neoadjuvant therapy

INTERVENTIONS:
Combination Product: neoadjuvant therapy — The enrolled patients undergo 2 cycles of neoadjuvant therapy, with each cycle consisting of treatment every 3 weeks. On the first day of the first treatment cycle, conventional transarterial chemoembolization (TACE) is performed, and concomitant intravenous infusion of tislelizumab at a dose of 200mg is given, followed by oral administration of lenvatinib at a dose of 8/12mg once daily. On the first day of the second cycle, tislelizumab is again administered intravenously at a dose of 200mg, TACE is not repeated, and lenvatinib treatment is continued. Within 2-4 weeks after the completion of neoadjuvant therapy, the investigator evaluates the tumor's suitability for surgical resection based on a comprehensive assessment of imaging results. Subsequently, eligible patients undergo tumor resection surgery, followed by follow-up for survival and safety monitoring.

SUMMARY:
In order to improve the R0 resection rate, reduce distant metastasis, and lower postoperative recurrence, there is a growing exploration of surgical treatments for hepatocellular carcinoma (HCC), including preoperative neoadjuvant therapy and postoperative adjuvant therapy. This study is a single-arm, prospective, exploratory clinical trial aimed at evaluating the effectiveness and safety of combining tislelizumab with transarterial chemoembolization (TACE) and lenvatinib as neoadjuvant therapy for resectable CNLC stage IIa-IIb HCC patients. The primary research endpoint of this study is recurrence-free survival (RFS). A total of 20 Chinese HCC patients with stage IIa-IIb and tumors deemed resectable by the investigator are enrolled in this study. For stage IIa patients, the inclusion criteria require meeting any of the following: unclear tumor boundaries, proximity to blood vessels, or suspicious residual margins. The enrolled patients undergo 2 cycles of neoadjuvant therapy, with each cycle consisting of treatment every 3 weeks. On the first day of the first treatment cycle, conventional transarterial chemoembolization (TACE) is performed, and concomitant intravenous infusion of tislelizumab at a dose of 200mg is given, followed by oral administration of lenvatinib at a dose of 8/12mg once daily. On the first day of the second cycle, tislelizumab is again administered intravenously at a dose of 200mg, TACE is not repeated, and lenvatinib treatment is continued. Within 2-4 weeks after the completion of neoadjuvant therapy, the investigator evaluates the tumor's suitability for surgical resection based on comprehensive assessment of imaging results. Subsequently, tumor resection surgery is performed on eligible patients, followed by survival and safety follow-up for the patients.

DETAILED DESCRIPTION:
1. Background

   Primary liver cancer is one of the most common malignancies worldwide, ranking sixth in terms of incidence and third in terms of cancer-related mortality. Hepatocellular carcinoma (HCC) is the predominant type of primary liver cancer, accounting for 85%-90% of cases. Treatment options for HCC include hepatectomy, transplantation, local ablation therapy, transarterial chemoembolization (TACE), radiation therapy, and systemic therapy. Hepatectomy is currently the preferred treatment for HCC, but the five-year recurrence rate after surgery is high, and the overall survival rate for early-stage HCC is relatively low. Therefore, improving the prognosis of HCC is of utmost importance.

   In recent years, there has been increasing exploration of surgical treatments for HCC, including neoadjuvant therapy and adjuvant therapy, to increase the R0 resection rate, reduce distant metastasis, and lower the risk of postoperative recurrence. Neoadjuvant therapy for HCC refers to interventions such as preoperative radiotherapy, interventional therapy, targeted therapy, immunotherapy, and portal vein embolization (PVE) administered to patients with resectable HCC who have a high risk of recurrence. These interventions aim to reduce liver inflammation, shrink tumors, and eliminate early-stage microlesions, thereby improving the curative resection rate and overall survival rate.

   However, there is limited research supporting neoadjuvant therapy for HCC, and its role in HCC treatment remains unclear. Neoadjuvant therapy has shown preliminary efficacy in various cancers, such as increasing resection rates and preserving sphincter function in colorectal cancer, demonstrating significant effects in early-stage non-small cell lung cancer and advanced malignant melanoma, and showing promise in resectable pancreatic cancer with high-risk factors. Previous explorations of neoadjuvant therapy for HCC have included hepatic artery chemotherapy, radiation therapy, and systemic therapy.

   With the emergence of immunotherapy and its promising efficacy in advanced liver cancer, research on immunotherapy as a neoadjuvant treatment has been conducted. Studies have shown that neoadjuvant treatment with immunotherapy in resectable liver cancer has achieved significant tumor necrosis and complete pathological responses. However, current clinical trials have not reached definitive conclusions, and the role of neoadjuvant therapy in patients with resectable HCC remains controversial. Therefore, this study aims to evaluate the efficacy and safety of Tislelizumab in combination with Transarterial Chemoembolization (TACE) and Lenvatinib as neoadjuvant therapy for patients with resectable CNLC stage IIa-IIb hepatocellular carcinoma (HCC), with the goal of providing a better treatment strategy to improve the survival outcomes of these patients.
2. Study Objectives

   2.1 Primary Objective:

   - To evaluate the recurrence-free survival (RFS) of patients with resectable CNLC stage IIa-IIb hepatocellular carcinoma (HCC) treated with Tislelizumab in combination with Transarterial Chemoembolization (TACE) and Lenvatinib as neoadjuvant therapy.

   2.2 Secondary Objectives:
   * To evaluate the objective response rate (ORR) of patients with resectable CNLC stage IIa-IIb HCC treated with Tislelizumab in combination with TACE and Lenvatinib as neoadjuvant therapy.
   * To evaluate the pathological complete response (pCR) rate of patients with resectable CNLC stage IIa-IIb HCC treated with Tislelizumab in combination with TACE and Lenvatinib as neoadjuvant therapy.
   * To evaluate the major pathological response (MPR) rate of patients with resectable CNLC stage IIa-IIb HCC treated with Tislelizumab in combination with TACE and Lenvatinib as neoadjuvant therapy.
   * To evaluate the R0 resection rates of patients with resectable CNLC stage IIa-IIb HCC treated with Tislelizumab in combination with TACE and Lenvatinib as neoadjuvant therapy.
   * To evaluate the overall survival (OS) of patients with resectable CNLC stage IIa-IIb HCC treated with Tislelizumab in combination with TACE and Lenvatinib as neoadjuvant therapy.
   * To assess the safety (according to NCI-CTCAE v5.0) of patients with resectable CNLC stage IIa-IIb HCC treated with Tislelizumab in combination with TACE and Lenvatinib as neoadjuvant therapy.
3. Study Design

   This is a single-arm, prospective, exploratory clinical trial aimed at investigating the effectiveness and safety of Tislelizumab combined with Transarterial Chemoembolization (TACE) and Lenvatinib as neoadjuvant therapy in approximately 20 patients with resectable CNLC stage IIa-IIb hepatocellular carcinoma (HCC) who have not received any prior treatment. Patients in CNLC stage IIa must meet one of the following criteria: unclear tumor margins, proximity to blood vessels, or suspicious residual margins. The primary endpoint of this study is recurrence-free survival (RFS), which will be assessed by the investigators based on the intention-to-treat (ITT) population assessment.

   Every effort will be made to ensure that the required tests and procedures outlined in the protocol are conducted according to plan. However, unforeseen circumstances may arise that are beyond the control of the investigators, making it difficult to perform the required assessments. In such cases, the investigators will take all necessary measures to ensure the safety and well-being of the participants. If a required assessment cannot be performed as specified in the protocol, the investigators will document the reasons for this occurrence. Additionally, any unexpected situations that occur will be promptly reported to the research team.

   3.1 Screening Period

   The investigators will enroll participants according to the following steps:

   3.1.1 Obtain informed consent with the participant's signature before conducting any study-related procedures.

   3.1.2 The principal investigator or designated personnel, who have undergone appropriate training, will review the inclusion/exclusion criteria to formally determine the eligibility of participants.

   3.2 Treatment Period

   During the treatment period, relevant physical examinations, laboratory tests, and collection of adverse events (AEs) and concomitant medication information will be conducted. The dispensing, retrieval, and inventory of medications will also be recorded.

   3.2.1 Neoadjuvant Stage
   * Tislelizumab: 200 mg, administered intravenously on the first day of each treatment cycle. Each cycle lasts for 3 weeks, with a total of 2 treatment cycles. The initial infusion (first day of the first cycle) should be completed within 60 minutes. If the infusion is well tolerated, subsequent infusions can be administered within 30 minutes, followed by an additional 2-hour patient monitoring period.
   * Lenvatinib: 8 mg per dose (for weight <60 kg) or 12 mg per dose (for weight ≥60 kg), taken orally once daily until one week before surgery. The medication should be taken at the same fixed time each day, with or without food. The tablets should be swallowed whole. Alternatively, the tablet (without opening or crushing it) can be mixed with one tablespoon of water or apple juice in a glass to form a suspension. If a dose is missed and cannot be taken within 12 hours, it should be skipped, and the next dose should be taken at the regular scheduled time.
   * TACE: One session of TACE will be performed on the first day of the neoadjuvant treatment, within the first cycle. The conventional TACE (cTACE) technique will be used in this study.

   3.2.2 Surgical Stage

   After completing the neoadjuvant treatment, the feasibility of surgery will be assessed by the investigator. Surgery will be performed for tumor resection within 2-4 weeks after the neoadjuvant treatment. The investigator and pathology department will conduct an assessment of neoadjuvant treatment response (MPR and pCR).

   3.2.3 Postoperative Stage

   After the final treatment, patients will enter the treatment follow-up and safety monitoring period. Patients who discontinue treatment due to disease progression should continue to be followed up for their survival. Patients who discontinue treatment or exit the study for reasons other than disease progression will undergo tumor assessment every 12 weeks until disease progression, death, study completion, or intolerable toxicity. The investigator may collect information on the patient's survival (date of death and cause of death) and other anti-tumor treatments after the completion of the study by conducting telephone interviews with the patient, their family members, or local physicians. The details of each survival follow-up should be accurately recorded in the original medical records. Safety follow-up is required for all patients within 90 days after the last treatment.
4. Efficacy and Safety Assessment

The ITT population includes all enrolled patients and serves as the primary analysis population for efficacy. The safety population includes all patients who received at least one dose of the investigational drugs and will be used for safety analysis.

4.1 Efficacy Assessment

* Recurrence-Free Survival (RFS): The time from the first day of curative surgery to tumor recurrence or death from any cause.
* Objective Response Rate (ORR): The proportion of participants with the best overall response (BOR) of complete response (CR) or partial response (PR) assessed by the investigator according to RECIST v1.1 during the neoadjuvant stage.
* Pathological Complete Response Rate (pCR): The proportion of patients assessed by the investigator, after completion of neoadjuvant treatment, with no residual tumor cells in the resected tumor.
* Major Pathological Response Rate (MPR): The proportion of patients assessed by the investigator, after completion of neoadjuvant treatment, with ≤10% residual viable tumor cells in the resected tumor.
* R0 Resection Rate: The proportion of patients achieving R0 resection among all surgical patients.
* Overall Survival (OS): The time from the start of treatment to death from any cause.

4.2 Safety Assessment

Safety will be evaluated by monitoring and recording all adverse events (AEs) and serious adverse events (SAEs) in terms of their incidence and severity, graded according to NCI-CTCAE v5.0. Laboratory test results (such as hematology, clinical chemistry, urine analysis), vital signs, ECOG performance status, and physical examinations will also be used to assess safety. Descriptive statistics will be used to analyze all safety data in the safety population.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must voluntarily enroll in this study and provide signed informed consent.
2. Male or female patients between the ages of 18 and 75 years old.
3. Patients diagnosed with hepatocellular carcinoma (HCC) confirmed by histopathology or imaging.
4. Chinese liver cancer staging of IIa-IIb with hepatocellular carcinoma considered resectable by the investigator. For IIa-stage patients, they must meet at least one of the following criteria: unclear tumor margins, proximity to blood vessels, or suspicious residual margins.
5. At least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1) guidelines (measurable lesions with CT scan long diameter ≥ 10 mm or lymph node lesions with CT scan short diameter ≥ 15 mm, and no prior local treatment such as radiation or cryotherapy).
6. Child-Pugh liver function class A.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. No prior systemic treatment for HCC.
9. For HBsAg-positive patients, HBV-DNA < 200,000 IU/ml (106 copies/ml), and receiving routine antiviral therapy.
10. Expected survival of at least 3 months.
11. Normal major organ function, meeting the following criteria:

    * Hematology criteria:
    * Hemoglobin (HB) ≥ 90 g/L;
    * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L (1500/m3);
    * Platelet count (PLT) ≥ 75 × 109/L.
    * Biochemistry criteria:
    * Total bilirubin (TBIL) ≤ 2 × ULN;
    * ALT, ALP, and AST ≤ 5 × ULN;
    * Serum creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance (CrCl) ≥ 50 ml/min (calculated using the Cockcroft-Gault formula: CrCL (mL/min) = [(140 - age) × body weight (kg) × F] / (SCr(mg/dL) × 72). Where F=1 for males and F=0.85 for females; SCr=serum creatinine).
    * Coagulation function: International Normalized Ratio (INR) ≤ 2.3.
12. Blood pressure (BP) controlled with a maximum of 3 antihypertensive medications, defined as BP ≤ 150/90 mmHg at screening, and no changes in antihypertensive treatment within one week before Cycle 1/Day 1.
13. Doppler echocardiography: Left Ventricular Ejection Fraction (LVEF) ≥ lower limit of normal (50%).
14. Women of childbearing potential must use reliable contraceptive methods or undergo pregnancy testing (serum or urine) within 7 days before enrollment, with negative results, and agree to use appropriate contraceptive methods during the trial and for 8 weeks after the last dose of investigational drugs. For males, they must agree to use appropriate contraceptive methods during the trial and for 8 weeks after the last dose of investigational drugs or have undergone surgical sterilization.

Exclusion Criteria:

1. Extrahepatic metastasis of primary liver cancer.
2. Diffuse liver cancer with tumor burden ≥ 50% of liver volume; and/or macrovascular invasion of the portal vein classified as Type IV; and/or inferior vena cava tumor thrombosis.
3. Prior treatment with targeted immunotherapy agents, including but not limited to anti-PD-1, anti-PD-L1, or anti-cytotoxic T-lymphocyte-associated antigen 4 (anti-CTLA-4) antibodies.
4. Contraindications for Transarterial Chemoembolization (TACE) treatment.
5. Participation in other investigational drug trials within the past 4 weeks.
6. Medical history and comorbidities:1)Active, known, or suspected autoimmune diseases, including a history of allogeneic organ transplantation, allogeneic hematopoietic stem cell transplantation, HIV positive history, or acquired immunodeficiency syndrome (AIDS) history. 2)Severe cardiovascular diseases: Grade II or higher myocardial ischemia or myocardial infarction, poorly controlled arrhythmia; NYHA Class III-IV heart failure, or left ventricular ejection fraction (LVEF) < 50% based on echocardiography. 3)Active infections. 4)Known allergies to components of Tislelizumab or Lenvatinib. 5)History of substance abuse, alcoholism, or drug addiction.
7. Ineligibility as determined by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
recurrence-free survival (RFS) | up to 36 months
  The period of time from the first day of curative surgery until tumor recurrence or death from any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 10 weeks
  The proportion of participants assessed by the investigators based on RECIST v1.1 criteria, who achieve a best overall response (BOR) of complete response (CR) or partial response (PR) during the neoadjuvant treatment period.
Pathological Complete Response Rate (pCR) | 10 weeks
  The proportion of patients evaluated by the investigators after completion of neoadjuvant treatment, who have no residual tumor cells in the resected tumor.
Major Pathological Response Rate (MPR) | 10 weeks
  The proportion of patients assessed by the investigators after completion of neoadjuvant treatment, who have residual viable tumor cells of ≤10% in the resected tumor.
R0 Resection Rate | 10 weeks
  The proportion of patients who achieve R0 resection among all surgical patients.
Overall Survival (OS) | up to 36 months
  The time from the start of treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Zhibo, PhD, Principal Investigator — First Affiliated Hospital of Fujian Medical University
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No